CLINICAL TRIAL: NCT00731107
Title: XCEL Bladeless Trocar Versus Veress Needle: A Randomised Controlled Trial Comparing These Two Entry Techniques in Gynaecological Laparoscopic Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southern Health (Other)
Responsible Party: Dr Thomas Manley, Southern Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRM-001
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Laparoscopic Surgery
Keywords: Veress Needle; XCEL bladeless trocar; Laparoscopic entry techniques
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Veress Needle laparoscopic entry
  Interventions: Procedure: laparoscopic surgery
- 2 (Active Comparator): XCEL bladeless trocar laparoscopic entry
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — XCEL bladeless trocar laparoscopic entry
  Arms: 2
Procedure: laparoscopic surgery — Veress Needle laparoscopic entry
  Arms: 1

SUMMARY:
The method most commonly used to gain entry to the abdomen in laparoscopic surgery (minimally invasive surgery) amongst gynecologists is the Veress Needle. This needle is inserted, usually near the belly button, before adding gas to the abdomen. With a pressurised abdomen a sharp trocar is then inserted to hold the operating telescope.

The XCEL bladeless trocar is another method of inserting the operating telescope whereby you don't need to first introduce gas before the trocar. This trocar is widely used in laparoscopic surgery but it is uncommon to the field of gynecology.

This study will compare the two methods with regard to:

1. Time taken to enter the abdomen
2. The number of attempts taken to enter the abdomen
3. The impact of the time taken to enter compared to the whole operating time
4. The happiness that the surgeon has entered the abdomen before adding gas, on a scale of 1 to 5.

Patients will be recruited into the trial through the Monash Medical Centre Gynecology department and the Mercy Hospital for Women Gynecology department. Patients that are having laparoscopic surgery and would usually have a Veress Needle entry are suitable for this trial. A patient information sheet will be provided and written consent will then be obtained. Patients who give written consent will be randomised into one of two arms of the trial, either the control (Veress Needle) or the XCEL bladeless trocar arm.

Information will be entered on a proforma by a researcher for each patient during their operation. All patient information will be strictly confidential and only be available to researchers directly involved in the study.

Surgeons operating as part of the project are the consultants and fellow of the gynecology department of Monash Medical Centre and Mercy Hospital for Women and are competent in both techniques.

200 women will be recruited over a one year period and the data will then be analysed with the help of a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Any woman having a Veress Needle laparoscopy through the Southern Health and Mercy Hospital for Women gynecology departments

Exclusion Criteria:

* Any women considered not eligible for a Veress Needle laparoscopy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Primary out come measure is time to entry in laparoscopic surgery | 1 year

SECONDARY OUTCOMES:
number of attempts at entry in laparoscopic surgery | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Health Department of Obstetrics and Gynaecology, Level 5, Monash Medical Centre, 256 Clayton Road, Clayton, Victoria, Australia